CLINICAL TRIAL: NCT05652114
Title: Examining the Impact of Mightier Play on Common Pediatric Symptoms in an Uncontrolled Environment
Brief Title: Open Label Mightier Play in the Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neuromotion Labs (Industry)
Responsible Party: Principal Investigator, Alyssa Peechatka, Lead Scientist, Neuromotion Labs
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NML
Record Dates: First submitted 2022-12-07; First posted 2022-12-15 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Emotional Regulation
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Intervention Model Description: As a single arm study all participants' children will receive a game-based biofeedback intervention. They are encouraged to engage with the intervention in an entirely self-directed manner.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Child play of Mightier (Experimental): Ad lib child biofeedback video game play in home
  Interventions: Behavioral: Mightier

INTERVENTIONS:
Behavioral: Mightier — Mightier is an app-based biofeedback video game that utilizes heart rate (HR) monitoring during game play to teach and facilitate practice of emotional regulation skills in children.

SUMMARY:
Mightier is a digital mental health tool that uses video game-based heart rate biofeedback to teach emotion regulation. The primary goal of this study is to replicate results from original clinical trials, demonstrating that playing Mightier at home improves common symptoms associated with emotional dysregulation.

Participants will be caregivers of children who are using Mightier, a video-game based heart rate biofeedback intervention. Caregivers will be asked to complete a short survey about their child's emotions and behaviors prior to their child's first play and then complete that survey two more times, at 8 weeks and 12 weeks post baseline.

The pre-post self report design will allow us to observe changes during Mightier use and relate those changes to overall engagement with the intervention

DETAILED DESCRIPTION:
Mightier is a video-game-based biofeedback intervention that capitalizes on children's love of video games to increase emotional awareness and facilitate emotion regulation practice through heart rate (HR) control. Each family receives a Mightier Kit (Mighty Band heart rate monitor and dedicated tablet), the Mightier App, online caregiver resources, and dedicated 1-on-1 support from a licensed clinician. The effectiveness of Mightier has been supported through several studies in children ages 8-18, specifically reducing symptoms of aggression, oppositional behavior, and parental stress. The core hypothesis underlying Mightier is that learning to regulate autonomic arousal via HR regulation during gameplay will lead to greater emotional regulation capacity. This hypothesis has considerable support, as greater dynamic HR control is associated with greater emotional clarity, emotion regulation, and impulse control in both adults and children.

Although originally created and studied in an academic medical center, it is not well understood how these learnings translate to change in a more diverse population in a less well-controlled environment (i.e. the home) with varying engagement with the intervention. Increased understanding of the Mightier population's behavioral and symptom characteristics, and the interplay between individual characteristics, engagement, HR, and symptom change is imperative to improving the intervention.

For this proposed study, we hypothesize the following:

1. Participants will report reduction in symptoms after 12 weeks of Mightier
2. Participants will show reduction in median HR during gameplay after 12 weeks of Mightier

   a. The magnitude of this change will be greater in externalizing symptoms
3. Change in symptoms will be inversely associated with total playtime such that children who play Mightier more will see the largest change (i.e. reduction) in symptoms
4. Changes in symptoms will be associated with change in median HR during gameplay, such that larger reductions in symptoms will be associated with larger reductions in HR during gameplay

After consent is obtained, caregivers will begin the survey. They will first be asked to identify whether symptoms associated with Anxiety, Attention Deficit Hyperactivity Disorder (ADHD), irritability, or aggression best describe their child. Based on these responses, caregivers will be asked to complete one of four validated symptom questionnaires. Those who indicated symptoms of anxiety best describe their child will complete the SCARED, a 41 item measure of symptoms of Anxiety related disorders. Those who indicated symptoms of ADHD best describe their child will complete the NICHQ Vanderbilt Assessment Scale, a 55 item measure of symptoms and ratings of functional performance associated with ADHD and Oppositional Defiant Disorder. Those who indicated aggression and aggressive behaviors best describe their child will complete the MOAS, a 4 item measure of verbal aggression, physical aggression, aggression against property, and autoaggression. Finally, those who indicated that symptoms of irritability best describe their child will complete the ARI a 7 item measure of irritability. Upon completion of the respective scale, caretakers will be thanked and informed that they will be contacted in approximately 8-12 weeks.

For the duration of the 8-12 week intervention period, participants will play Mightier ad libitum.

ELIGIBILITY:
Inclusion Criteria:

* Parent or caregivers have a child engaging with the heart rate biofeedback intervention Mightier

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2732 (Actual)
Dates: Start 2020-04-10 (Actual); Primary Completion 2022-11-17 (Actual); Study Completion 2022-11-17 (Actual)

PRIMARY OUTCOMES:
Affective Reactivity Index - Parent | 12 weeks
  The Affective Reactivity Index is a 7 item parent reported measure of irritability. Scores range from 0-12, with higher scores representing greater irritability.
Modified Overt Aggression Scale | 12 weeks
  The Modified Overt Aggression Scale is a 4 item, caregiver report measure of verbal aggression, physical aggression, aggression against property, and autoaggression. Scores range from 0 to 40, with higher scores indicating more aggression.

SECONDARY OUTCOMES:
Screen for Anxiety Related Emotional Disorders | 12 weeks
  The Screen for Anxiety Related Emotional Disorders is a 41 item measure of symptoms of anxiety related disorders. Scores range from 0-82, with higher scores representing more severe anxiety. Scores >25 indicating high likelihood of an anxiety disorder.
National Institute for Children's Health Quality Vanderbilt Assessment Scale | 12 weeks
  NIHQ Vanderbilt Assessment Scale is a 55 item measure of symptoms and ratings of functional performance associated with ADHD and Oppositional Defiant Disorder. Scores are broken into 5 subscales with a set of performance questions. Higher scores on all scales represent more severe symptoms and/or impairment. To meet criteria across all 5 domains, parents must endorse a score of 2 or 3 on a specified number of symptoms and a 4 or 5 on at least one performance question.

CONTACTS AND LOCATIONS:
Locations (1):
- Neuromotion Inc, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No